CLINICAL TRIAL: NCT03722927
Title: The Use of Liposomal Bupivacaine for Pain Control Following Mastectomy and Breast Reconstruction
Brief Title: The Use Of Liposomal Bupivacaine For Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00045562
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2021-05

CONDITIONS: Pain, Breast
Keywords: Bupivacaine; Liposomal Bupivacaine; Mastectomy; Breast Reconstruction; Pain Control
MeSH Terms: conditions — Mastodynia; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Women of all races and ethnicity who meet the above-described eligibility criteria are eligible to participate in this study. Approximately 5% of study participants to be Hispanic/Latino (N=5), 10% Black or African American (N=10), 1% American Indian/Alaska Native (N=1), and 5% Asian (N=5).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine Group (Experimental): Participants will be randomized to the Bupivacaine Group and receive a bilateral mastectomy with immediate implant based breast reconstruction
  Interventions: Drug: Bupivacaine
- Liposomal Bupivacaine Group (Experimental): Participants will be randomized to the Liposomal Bupivacaine Group and receive a bilateral mastectomy with immediate implant based breast reconstruction
  Interventions: Drug: Liposomal Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — While in the operating room,if subject is randomized to bupivacaine, it will be injected into the surgical site. After surgery, oral and IV pain medications will be available to control pain. During the hospital stay, subject will rate pain on pain scales and monitor how much pain medications needed. Once discharged, PI/staff will provide a pain diary to record pain medication use and pain rating (0-10). Subjects will follow up with clinic at regularly scheduled appointment times at 1 week, 3 weeks and 5 weeks postoperatively. At those appointments, PI/staff will have subjects bring pain medication diary and fill out a pain assessment and a disability assessment related to recent surgery.
  Other Names: Marcaine
  Arms: Bupivacaine Group
Drug: Liposomal Bupivacaine — While in the operating room,if subject is randomized to Liposomal Bupivacaine, it will be injected into the surgical site. After surgery, oral and IV pain medications will be available to control pain. During the hospital stay, subject will rate pain on pain scales and monitor how much pain medications needed. Once discharged, PI/staff will provide a pain diary to record pain medication use and pain rating (0-10). Subjects will follow up with clinic at regularly scheduled appointment times at 1 week, 3 weeks and 5 weeks postoperatively. At those appointments, PI/staff will have subjects bring pain medication diary and fill out a pain assessment and a disability assessment related to recent surgery.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine Group

SUMMARY:
The purpose of this research study is to determine how well the local anesthetic, liposomal bupivacaine, controls postoperative pain after mastectomy and breast reconstruction.

DETAILED DESCRIPTION:
Eligible subjects will be identified prior to surgery. On the day of surgery, each patient will be randomized to be in either Local infiltration of bupivacaine OR liposomal bupivacaine. Study will be double blinded to patients and Investigators. Patients assigned to the local infiltration with bupivacaine group will receive a total 60 ml of 0.25% bupivacaine with 30 ml delivered to each breast. Patients assigned to the local infiltration of liposomal bupivacaine will receive a total of 20 ml liposomal bupivacaine (266 mg) with 10 ml of 0.25% bupivacaine and 30 ml of 0.9% sodium chloride. These injections will occur at the end of the mastectomy and prior to the insertion of the tissue expander implant. After this intraoperative injection, patients will not receive any more doses of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive a bilateral mastectomy with immediate sub-pectoral implant based breast reconstruction
* Age ≥ 18 years
* Ability to understand and the willingness to sign an (Institutional Review Board) IRB-approved informed consent document.
* Patients who receive tissue expander placement or direct permanent implant placement will be included in the study.

Exclusion Criteria:

* Patients who receive an autologous tissue reconstruction.
* Patients who receive a unilateral reconstruction.
* Patients who are expected to undergo axillary lymph node dissection
* Patients who have undergone breast irradiation
* Patients who abuse narcotics or have chronic pain (using greater than 40 mg equivalents of oxycodone per day)
* Patients who are wards of the state
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bupivacaine or liposomal bupivacaine.
* Pregnant women are excluded from this study because pregnancy precluded immediate breast reconstruction in our patient population.
* Patients who weigh less than 50 kg, as there can be dose related toxicities of the bupivacaine dosing used n this study.
* Patients with moderate-severe hepatic or renal impairment because of the increased risk of toxicity.
* Patients receiving bilateral mastectomy with immediate pre-pectoral implant based reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Runyan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Lovecchio F, Jordan SW, Lim S, Fine NA, Kim JY. Risk Factors for Complications Differ Between Stages of Tissue-Expander Breast Reconstruction. Ann Plast Surg. 2015 Sep;75(3):275-80. doi: 10.1097/SAP.0000000000000109. PMID 24691330
- [Background] Butz DR, Shenaq DS, Rundell VL, Kepler B, Liederbach E, Thiel J, Pesce C, Murphy GS, Sisco M, Howard MA. Postoperative Pain and Length of Stay Lowered by Use of Exparel in Immediate, Implant-Based Breast Reconstruction. Plast Reconstr Surg Glob Open. 2015 Jun 5;3(5):e391. doi: 10.1097/GOX.0000000000000355. eCollection 2015 May. PMID 26090281
- [Background] Ng SK, Hare RM, Kuang RJ, Smith KM, Brown BJ, Hunter-Smith DJ. Breast Reconstruction Post Mastectomy: Patient Satisfaction and Decision Making. Ann Plast Surg. 2016 Jun;76(6):640-4. doi: 10.1097/SAP.0000000000000242. PMID 25003439
- [Background] Shekhawat L, Busheri L, Dixit S, Patel C, Dhar U, Koppiker C. Patient-Reported Outcomes Following Breast Reconstruction Surgery and Therapeutic Mammoplasty: Prospective Evaluation 1 Year Post-Surgery with BREAST-Q Questionnaire. Indian J Surg Oncol. 2015 Dec;6(4):356-62. doi: 10.1007/s13193-015-0432-x. Epub 2015 Jul 23. PMID 27065661
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Morrison JE Jr, Jacobs VR. Reduction or elimination of postoperative pain medication after mastectomy through use of a temporarily placed local anesthetic pump vs. control group. Zentralbl Gynakol. 2003 Jan;125(1):17-22. doi: 10.1055/s-2003-40364. PMID 12877104
- [Background] Lee MJ, Daniels SL, Wild JRL, Wilson TR; SYSuRG RAGeS Group. Readmissions after general surgery: a prospective multicenter audit. J Surg Res. 2017 Mar;209:53-59. doi: 10.1016/j.jss.2016.09.020. Epub 2016 Sep 19. PMID 28032571
- [Background] Bonnet F, Marret E. Influence of anaesthetic and analgesic techniques on outcome after surgery. Br J Anaesth. 2005 Jul;95(1):52-8. doi: 10.1093/bja/aei038. Epub 2004 Dec 3. PMID 15579487
- [Background] Strang P. Cancer pain--a provoker of emotional, social and existential distress. Acta Oncol. 1998;37(7-8):641-4. doi: 10.1080/028418698429973. PMID 10050980
- [Background] Zielinski T, Lorenc-Podgorska K, Antoszewski B. Why women who have mastectomy decide not to have breast reconstruction? Pol Przegl Chir. 2015 Feb 3;86(10):451-5. doi: 10.2478/pjs-2014-0081. PMID 25720103
- [Background] American Society of Plastic Surgeons. (2015). Plastic surgery statistics report. Retrived from https://d2wirczt3b6wjm.cloudfront.net/News/Statistics/2015/plastic-surgery-statistics-full-report-2015.pdf
- [Background] Gassman AA, Yoon AP, Festekjian J, Da Lio AL, Tseng CY, Crisera C. Comparison of immediate postoperative pain in implant-based breast reconstructions. J Plast Reconstr Aesthet Surg. 2016 May;69(5):604-16. doi: 10.1016/j.bjps.2015.12.009. Epub 2016 Jan 7. PMID 26947947
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- [Background] Viscusi ER, Sinatra R, Onel E, Ramamoorthy SL. The safety of liposome bupivacaine, a novel local analgesic formulation. Clin J Pain. 2014 Feb;30(2):102-10. doi: 10.1097/AJP.0b013e318288e1f6. PMID 23446090
- [Background] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Background] Fayezizadeh M, Majumder A, Neupane R, Elliott HL, Novitsky YW. Efficacy of transversus abdominis plane block with liposomal bupivacaine during open abdominal wall reconstruction. Am J Surg. 2016 Sep;212(3):399-405. doi: 10.1016/j.amjsurg.2015.12.026. Epub 2016 Apr 12. PMID 27156796
- [Background] Rawlani V, Kryger ZB, Lu L, Fine NA. A local anesthetic pump reduces postoperative pain and narcotic and antiemetic use in breast reconstruction surgery: a randomized controlled trial. Plast Reconstr Surg. 2008 Jul;122(1):39-52. doi: 10.1097/PRS.0b013e3181774349. PMID 18594373
- [Background] Nadeau MH, Saraswat A, Vasko A, Elliott JO, Vasko SD. Bupivacaine Versus Liposomal Bupivacaine for Postoperative Pain Control after Augmentation Mammaplasty: A Prospective, Randomized, Double-Blind Trial. Aesthet Surg J. 2016 Feb;36(2):NP47-52. doi: 10.1093/asj/sjv149. Epub 2015 Dec 23. PMID 26704270
- [Background] Smoot JD, Bergese SD, Onel E, Williams HT, Hedden W. The efficacy and safety of DepoFoam bupivacaine in patients undergoing bilateral, cosmetic, submuscular augmentation mammaplasty: a randomized, double-blind, active-control study. Aesthet Surg J. 2012 Jan;32(1):69-76. doi: 10.1177/1090820X11430831. Epub 2011 Dec 16. PMID 22179931
- [Background] Coopey SB, Specht MC, Warren L, Smith BL, Winograd JM, Fleischmann K. Use of preoperative paravertebral block decreases length of stay in patients undergoing mastectomy plus immediate reconstruction. Ann Surg Oncol. 2013 Apr;20(4):1282-6. doi: 10.1245/s10434-012-2678-7. Epub 2012 Oct 14. PMID 23064793
- [Background] Andersen KG, Christensen KB, Kehlet H, Bidstup PE. The Effect of Pain on Physical Functioning After Breast Cancer Treatment: Development and Validation of an Assessment Tool. Clin J Pain. 2015 Sep;31(9):794-802. doi: 10.1097/AJP.0000000000000156. PMID 25679946
- [Background] Campbell I, Cavanagh S, Creighton J, French R, Banerjee S, Kerr E, Shirley R. To infiltrate or not? Acute effects of local anaesthetic in breast surgery. ANZ J Surg. 2015 May;85(5):353-7. doi: 10.1111/ans.12541. Epub 2014 Apr 22. PMID 24754798
- [Background] Byager N, Hansen MS, Mathiesen O, Dahl JB. The analgesic effect of wound infiltration with local anaesthetics after breast surgery: a qualitative systematic review. Acta Anaesthesiol Scand. 2014 Apr;58(4):402-10. doi: 10.1111/aas.12287. PMID 24617619
- [Background] Zielinski J, Jaworski R, Smietanska I, Irga N, Wujtewicz M, Jaskiewicz J. A randomized, double-blind, placebo-controlled trial of preemptive analgesia with bupivacaine in patients undergoing mastectomy for carcinoma of the breast. Med Sci Monit. 2011 Oct;17(10):CR589-97. doi: 10.12659/msm.881986. PMID 21959614
- [Background] Tam KW, Chen SY, Huang TW, Lin CC, Su CM, Li CL, Ho YS, Wang WY, Wu CH. Effect of wound infiltration with ropivacaine or bupivacaine analgesia in breast cancer surgery: A meta-analysis of randomized controlled trials. Int J Surg. 2015 Oct;22:79-85. doi: 10.1016/j.ijsu.2015.07.715. Epub 2015 Aug 12. PMID 26277531
- [Background] US Food and Drug Administration. FDA Label Approved on 10/28/2011 for Exparel. US Silver Spring, MD: US Food and Drug Administration. Available from: http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/022496s000lbl.pdf
- [Background] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] US Food and Drug Administration. Marcaine Bupivcacaine HCl Injection Label. US Silver Spring, MD: US Food and Drug Administration. Available from: https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/018692s015lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 54 [54 to 54] | 48 [44 to 53] | 50 [44 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Analog Scores
Description: This will be measured every 12 hours for the first 48 hours postoperatively by the level of breast pain associated with arm movements while eating on a scale of 0-10 with higher scores denoting worse outcomes.
Time Frame: 48 hours
Population: Data was not collected for participant in the Bupicaine group at 24, 36 and 48 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 1 | 2
score on a scale
  12 hours | 4 [4 to 4] | 3.5 [3 to 4]
  24 hours: number analyzed (Participants) | 0 | 2
  24 hours |  | 4 [2 to 6]
  36 hours: number analyzed (Participants) | 0 | 2
  36 hours |  | 3.5 [3 to 4]
  48 hours: number analyzed (Participants) | 0 | 2
  48 hours |  | 2 [2 to 2]

2. Secondary Outcome: Area Under the Curve Visual Analog Scores (Submuscular Augmentation Mammoplasty)
Description: This will be measured during first 48 hours postoperatively
Time Frame: 48 hours
Population: Unable to calculate, data not collected at 48hours for Bupivacaine group or Liposomal Bupivacaine Group.
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Morphine Doses Across All Subjects
Description: This will be measured by the number of doses within the first month postoperatively and recorded on pain medication daily diary kept by subject.
Time Frame: 1 Month
Measure: Number; unit: Number of morphine doses
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 1 | 2
Number of morphine doses | 0 | 20

4. Secondary Outcome: Length of Stay for Hospitalization
Description: The length of stay for hospitalization after mastectomy and breast reconstruction will be recorded.
Time Frame: up to 47 Hours
Measure: Mean (Full Range); unit: days
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 1 | 2
days | 1 [1 to 1] | 1 [1 to 1]

5. Secondary Outcome: Readmission Rates to the Hospital
Description: Readmission rates to the hospital within 2 months after mastectomy and breast reconstruction will be recorded
Time Frame: Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

6. Secondary Outcome: Frequency of Postoperative Opioid Related Adverse Effects
Description: Frequency of postoperative opioid related adverse effects within the first week of surgery will be recorded. This includes nausea, vomiting, pruritus, allergy, respiratory depression.
Time Frame: Postoperatively, 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

7. Secondary Outcome: Pain Intensity With Movement
Description: This will be measured by using the Pain Assessment Questionnaire. Total scores are 0-50 with higher scores denoting worse outcomes.
Time Frame: Up to 2 months
Population: Data not collected
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months after intervention
Arm/Group | Bupivacaine Group | Liposomal Bupivacaine Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03722927/Prot_SAP_002.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03722927/ICF_001.pdf